CLINICAL TRIAL: NCT03417141
Title: Valchlor in the Treatment of Lichen Planopilaris: A Single Arm, Open- Label, Exploratory Study
Brief Title: Valchlor in the Treatment of Lichen Planopilaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Jason Sluzevich MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 16-006731
Record Dates: First submitted 2018-01-08; First posted 2018-01-31 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Lichen Planopilaris
Keywords: Valchor
MeSH Terms: conditions — Lichen Planus | interventions — Mechlorethamine; Amines

STUDY DESIGN:
Intervention Model Description: Adults patient with active Lichen Planopilaris or Frontal Fibrosing Alopecia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valchor treatment of Lichen Planopilaris (Experimental): Once daily application of Valchlor in decreasing disease activity in patients with Lichen Planopilaris.
  Interventions: Drug: Mechlorethamine 0.016% Top Gel

INTERVENTIONS:
Drug: Mechlorethamine 0.016% Top Gel — Valchlor, a 0.016% gel formulation of mechlorethamine. Once daily application of Valchlor in decreasing disease activity in patients with Lichen Planopilaris.
  Other Names: Valchlor

SUMMARY:
The primary objective of this study is to assess the potential effectiveness of once daily application of Valchlor in decreasing disease activity in patients with Lichen Planopilaris. The primary measurement of efficacy will be with the Lichen Planopilaris Activity Index (LPPAI) before and after 6 months of treatment. Secondary measures of efficacy will be the mean follicular density, Physician Global assessment (PGA) score, and the Dermatology Quality of Life Index (DQLI) score before and after six months of therapy.

DETAILED DESCRIPTION:
This is a single arm, open label, exploratory study to evaluate the efficacy of Valchlor in the treatment of LPP. Subjects will be screened by the Department of Dermatology at the Mayo Clinic in Florida outpatient clinic and interested qualified subjects will be consented and offered participation. This study is designed to establish feasibility and proof of concept and will not include randomization or crossover components.

Patients with biopsy proven LPP who have failed one prior topical or systemic therapy with evidence of active disease will be eligible to participate. The presence of active disease will be based on a baseline clinical exam showing perifollicular erythema with scaling. Patients with predominance of end stage scarring hair loss but without significant active erythema will be excluded. Involvement restricted to the frontal scalp is a recognized clinical variant of LPP and is known as frontal fibrosing alopecia (FAA). As the histological features of LPP and FAA are identical, patients with FAA subtype of LPP would also be eligible to participate in the study.

Eligible participants using high-potency topical corticosteroids, intralesional corticosteroids, or oral hydroxychloroquine may enroll but will be required to discontinue use during the study period.

All study participants will apply Valchlor 0.016% gel to involved areas at night. Patients will be instructed to first part the hair away from involved area as needed, limit application to areas with alopecia and erythema, apply 30 minutes after showering or washing, and allow treated areas to dry for 5 to 10 minutes before covering with clothing or going to bed. Participants will be instructed to wash their hands with soap and water after applying Valchlor. Caregivers who assist in application will be instruction to wear disposable nitrile gloves when applying Valchlor and dispose with the household trash. Patients will be instructed to store Valchlor in the refrigerator away from foods at 36°F - 46°F and apply within 30 minutes after removing from refrigeration.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years or older.
* Biopsy proven diagnosis of Lichen Planopilaris
* Biopsy proven diagnosis of Fontal Fibrosing Alopecia (a clinical variant of LPP restricted to frontal scalp)
* Good general health as confirmed by medical history
* Patients who are willing and capable of cooperating to the extent and degree required by the protocol; and
* Patients who read and sign an approved informed consent for this study

Exclusion Criteria:

* Vulnerable study population
* Pregnant or nursing women
* Women planning a pregnancy within the study period
* Active smokers
* Known history of adverse reaction to mechlorethamine
* Use of systemic immunosuppressive
* Presence of ulcerated scalp lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sluzevich, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Valchor Treatment of Lichen Planopilaris: Once daily application of Valchlor in decreasing disease activity in patients with Lichen Planopilaris.
  Valchlor: Valchlor, a 0.016% gel formulation of mechlorethamine. Once daily application of Valchlor in decreasing disease activity in patients with Lichen Planopilaris.
Period: Overall Study
Arm/Group | Valchor Treatment of Lichen Planopilaris
Started | 12
Completed | 8
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: All washed out prior treatments for 4 weeks before starting Valchor topically.
Arm/Group | Valchor Treatment of Lichen Planopilaris
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 66 [50 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12
LICHEN PLANOPILARIS ACTIVITY INDEX (LPPAI) [Median (Full Range); unit: Integer] — LPPAI index is a numeric score to quantify the signs and symptoms of LPP and frontal fibrosing alopecia (FFA) and records symptoms (pruritus, pain, burning), signs (erythema, perifollicular erythema and scale), a measure of activity (the anagen pull test), and extension of disease. Score ranges are from 0 to 10 on an integer scale. Higher scores represent more severe disease.
  Integer | 5 [3 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Change in Lichen Planopilaris Activity Index (LLPAI)
Description: The Lichen Planopilaris Activity Index is a standardized validated quantitative measure of disease activity. LPPAI score (0-10) is calculated as follows: (pruritus + pain + burning)/3 + (scalp erythema + perifollicular erythema + perifollicular scale)/3 + 2.5 (pull test) + 1.5 (spreading/2). Symptoms and signs are graded on a 4-point scale with 0 = absent, 1 = mild, 2 = moderate, and 3 =severe. Clinical progression and a positive hair pull test are graded 1=yes; 0=no. The percent change of LLPAI score from before and after treatment.
Time Frame: baseline, up to 24 weeks
Population: One subject withdrew and data was not analyzed for that subject
Measure: Median (Full Range); unit: percentage of change from baseline
Arm/Group | Valchor Treatment of Lichen Planopilaris
Number analyzed (Participants) | 11
percentage of change from baseline
  Week 12 | -42.9 [-100.0 to 33.3]
  Week 24 | -66.7 [-100.0 to 66.7]
Statistical Analysis 1: Comparison: Valchor Treatment of Lichen Planopilaris; Week 12; Test type: Superiority; p = 0.014, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Valchor Treatment of Lichen Planopilaris; Week 24; Test type: Superiority; p = 0.006, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Dermatology Quality of Life Index (DQLI)
Description: The DQLI is 10 standardized items measuring impact of skin disease rated as 0=not at all/not relevant; 1=a little; 2=a lot; 3=very much. The absolute change of total DQLI score from before and after treatment
Time Frame: baseline, 24 weeks
Population: One subject withdrew and three subjects were non-compliant with study procedures. Data was not analyzed for a total of four subjects.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Valchor Treatment of Lichen Planopilaris
Number analyzed (Participants) | 8
score on a scale | -2 [-11 to 2]
Statistical Analysis 1: Comparison: Valchor Treatment of Lichen Planopilaris; Test type: Superiority; p = 0.093, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Follicular Units
Description: Phototrichograms of all subjects scalps performed using FotoFinder video-epiluminescence microscopy (FotoFinder Systems GmbH) in combination with TrichoScan digital image analysis (TRICHOLOG GmbH and DatInf mbH). The percent change in the total number of hairs per square cm was measured before and after treatment.
Time Frame: baseline, 24 weeks
Population: One subject withdrew, and three subjects were non-compliant with study procedures. Data was not was not analyzed for a total of four subjects.
Measure: Median (Full Range); unit: percent change
Arm/Group | Valchor Treatment of Lichen Planopilaris
Number analyzed (Participants) | 8
percent change | -9.1 [-25.8 to 37.5]
Statistical Analysis 1: Comparison: Valchor Treatment of Lichen Planopilaris; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Mean Follicular Density
Description: Phototrichograms of all subjects scalps performed using FotoFinder video-epiluminescence microscopy (FotoFinder Systems GmbH) in combination with TrichoScan digital image analysis (TRICHOLOG GmbH and DatInf mbH). The percent change in the mean number of follicular units per square cm was measured before and after treatment.
Time Frame: baseline, 24 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: percent change
Arm/Group | Valchor Treatment of Lichen Planopilaris
Number analyzed (Participants) | 8
percent change | -9.0 [-25.8 to 37.6]
Statistical Analysis 1: Comparison: Valchor Treatment of Lichen Planopilaris; Test type: Superiority; p = 0.55, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collect for each subject from baseline until last treatment for a total of approximately six months
Arm/Group | Valchor Treatment of Lichen Planopilaris
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valchor Treatment of Lichen Planopilaris (N=12)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 11 (11)
Severe Itching (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
One subject withdrew and three subjects were non-compliant with study procedures. Data was not analyzed for a total of four subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03417141/Prot_SAP_000.pdf